CLINICAL TRIAL: NCT05426174
Title: Phase I, Randomized, Modified Double-blind, Parallel-group, Active-controlled, Multi-arm, Dose-escalation Study to Assess the Safety and Immunogenicity of Monovalent mRNA NA Vaccine in Adult Participants 18 Years of Age and Older
Brief Title: Study to Assess the Safety and Immunogenicity of Monovalent mRNA NA Vaccine in Adult Participants 18 Years of Age and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FBP00012; U1111-1266-5326 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-06-08; First posted 2022-06-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Influenza Immunization; Healthy Volunteers
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study will be blinded to participants, investigators/sub-investigators, outcomes assessors, laboratory personnel, and the sponsor study staff (with the exception noted for study staff involved in the ESDRs). Study staff involved in the ESDRs will be unblinded to group assignment of participants in the sentinel safety cohorts. After the ESDRs are performed for the sentinel safety cohorts, the SMT will continue monitoring the safety aspects of the study as part of blinded periodic safety reviews. Those preparing/administering the study interventions will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 mRNA NA: Low dose Level (Experimental): Participants will receive a low dose of mRNA vaccine
  Interventions: Biological: mRNA NA vaccine
- Group 2 mRNA NA: Medium dose level (Experimental): Participants will receive a medium dose of mRNA vaccine
  Interventions: Biological: mRNA NA vaccine
- Group 3 mRNA NA: High dose level (Experimental): Participants will receive a high dose of mRNA vaccine
  Interventions: Biological: mRNA NA vaccine
- Group 4: QIV-HD (Active Comparator): Participants will receive QIV-HD (high dose quadrivalent influenza) vaccine
  Interventions: Biological: High Dose Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: mRNA NA vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Group 1 mRNA NA: Low dose Level; Group 2 mRNA NA: Medium dose level; Group 3 mRNA NA: High dose level
Biological: High Dose Quadrivalent Influenza Vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Other Names: Fluzone HD
  Arms: Group 4: QIV-HD

SUMMARY:
This is a Phase I, first-in-human, randomized, modified double-blind, active-controlled, dose-escalation study to assess the safety and immunogenicity of up to 3 dose levels of mRNA NA vaccines, administered as a single IM injection in healthy adults aged 18 years and older. Two age groups, 18 to 64 years and ≥65 years, will be included in this study.

DETAILED DESCRIPTION:
This study will include a screening visit, 6 study visits occurring on Days 1, 3, 9, 29, 91, and 181, and a safety follow-up telephone call on Day 366.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older on the day of inclusion.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  1. Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile OR
  2. Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 12 weeks after study intervention administration
* A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 8 hours before administration of study intervention.
* Informed consent form has been signed and dated.

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the study intervention components; history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances
* Moderate or severe acute illness/infection (according to investigator judgement) or febrile illness (temperature ≥100.4°F) on the day of study intervention administration.
* Have known or recently active (12 months) neoplastic disease or a history of any hematologic malignancy.
* Have any diagnosis, current or past, of autoimmune disease.
* Body mass index of 40 kg/m2 or higher.
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Have taken high-dose inhaled corticosteroid (≥500 μg of fluticasone) within 6 months prior to study vaccination.
* Self-reported or documented seropositivity for HIV, hepatitis B virus, or hepatitis C virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events | Within 30 minutes after vaccination
  Immediate adverse events are unsolicited systemic adverse events reported in the 30 minutes after vaccination
Number of participants with solicited injection site or systemic reaction | From Day 1 to Day 8
Number of participants with unsolicited adverse events | From Day 1 to Day 29
  Unsolicited (spontaneously reported) adverse events not fulfilling criteria for solicited reactions
Number of participants with serious adverse events | From Day 1 to Day 366
  Serious adverse events are collected throughout the study
Number of participants with adverse events of special interest | From Day 1 to Day 366
  Adverse events of special interest are collected throughout the study
Number of patients with clinically significant changes in clinical laboratory tests | From Day 1 to Day 8
  Laboratory tests include hematology: complete blood count (CBC) with differential, platelet count, coagulation panel (prothrombin time and PTT) and serum chemistry: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total and fractionated bilirubin, C-reactive protein, serum creatinine, and blood urea nitrogen

SECONDARY OUTCOMES:
Neuraminidase inhibition (NAI) Antibodies at Day 1 and 29 | Day 1 and 29
  Antibody are expressed as GMTs at baseline and post-baseline
Individual Neuraminidase inhibition (NAI) titer | Day 1 and Day 29
  Antibody titers are expressed as GMTs at baseline and post-baseline
2-fold and 4-fold rise in NAI antibody titers | From Day 1 to Day 29
  Expressed as percentage post-baseline
Percentage of participants with detectable antibody titers greater than or equal to (≥) 10 [1/dil] | Day 1 and Day 29
  Expressed as percentage at baseline and post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- United States (6):
  - AES - DRS - Optimal Research_Site 8400007, Huntsville, Alabama
  - Central Phoenix Medical Clinic, LLC_Site: 8400010, Phoenix, Arizona
  - Optimal Research San Diego, LLC_Site: 8400009, San Diego, California
  - AES - DRS - Optimal Research_Site 8400002, Melbourne, Florida
  - AES - DRS - Optimal Research_Site 8400001, Peoria, Illinois
  - Synexus Clinical Research_Site 8400003, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: FBP00012 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25267&tenant=MT_SNY_9011